CLINICAL TRIAL: NCT01540591
Title: Does Intralipid Infusion Improve the Implantation Rate in Repeated Implantation Failure: a Randomized Controlled Trial
Brief Title: Intralipid for Repeated Implantation Failure
Acronym: Intralipid
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Waleed El-khayat, Assisstant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22012
Record Dates: First submitted 2012-02-23; First posted 2012-02-29 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Infertility
Keywords: repeated implantation failure; intralipid
MeSH Terms: conditions — Infertility | interventions — soybean oil, phospholipid emulsion; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control (Placebo Comparator): Saline 0.9% IV infusion between day 4 and 9 of ovarian stimulation & another dose when got pregnant within the 1st week of positive pregnancy test
  Interventions: Drug: Saline
- intralipid (Experimental): IV infusion of intralipid 20% between day4 and 9 of ovarian stimulation & another dose when got pregnant within the 1st week of positive pregnancy test
  Interventions: Drug: intralipid

INTERVENTIONS:
Drug: intralipid — IV infusion of intralipid 20% between day4 and 9 of ovarian stimulation & another dose when got pregnant within the 1st week of positive pregnancy test
  Other Names: intralipid 20%
  Arms: intralipid
Drug: Saline — Saline 0.9% IV infusion between day4 and 9 of ovarian stimulation & another dose when got pregnant within the 1st week of positive pregnancy test
  Other Names: Saline 0.9%
  Arms: control

SUMMARY:
Intralipid infusion can improve outcome in women with recurrent Intracytoplasmic sperm injection ( ICSI) failure due to elevated TH1 cytokine response.

DETAILED DESCRIPTION:
Infertile patients undergoing Intracytoplasmic Sperm Injection (ICSI) cycle with history of repeated implantation failure, intralipid will be given to the intervention group.

The primary outcome measure is the clinical pregnancy rate, secondary outcome measures implantation rate, ongoing pregnancy rate, abortion rate.

ELIGIBILITY:
Inclusion Criteria:

* Infertile patients undergoing ICSI cycle with history of repeated implantation failure

Exclusion Criteria:

1. Disturbances of normal fat metabolism such as pathologic hyperlipemia
2. Allergic to it; or to eggs, soybean oil, or safflower oil.
3. Severe liver disease, kidney disease, lung disease, anemia, blood clotting disorder.
4. Uterine fibroid, endometrial polyp, endometriosis and hydrosalpinx.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2012-02; Primary Completion 2013-09 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
clinical pregnancy rate | 10 month
  pregancy sac with fetal heart activity

SECONDARY OUTCOMES:
implantation rate | 10 month
  the number of gestational sacs divided by the number of embryos transferred
ongoing pregnancy rate | 14 month
  clinical pregnancy continue after 12 weeks gestational age

CONTACTS AND LOCATIONS:
Overall Officials: Waleed El-khayat, M.D., Principal Investigator — Faculty of medicine, Cairo University, Cairo, Egypt
Locations (1):
- Kasr Al-ainy hospital, Cairo, Egypt